CLINICAL TRIAL: NCT07089407
Title: Ten-Year Follow-Up Analysis of MBL and PES Outcomes Around Convergent Transmucosal Profile Implants
Brief Title: Ten Year Follow up of Convergent Profile Implants
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Associate Professor, University of Cagliari
Other Study IDs: Biotype retro
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Peri-implant Bone Loss; Peri-Implant Tissues
Keywords: Implants; Transmucosal profile; Marginal bone loss; Pink esthetic score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dental implant placement — Implant site prepared through a consecutive drilling procedure in the maxilla or the mandible, implant placed.

SUMMARY:
The aim of the study is to evaluate the marginal bone level (MBL) and pink aesthetic score (PES) changes on the short, medium and long-term, on a retrospective cohort of patients who received at least one "biotype implant" (DEI ITALIA SRL, Mercallo VA, Italy) with convergent transmucosal profile. Ninety-seven patients with at least one periapical x-ray taken on the day of implant placement and at least one taken in the following 10 years were included for MBL analysis and 90 patients who had at least one photograph taken on the day of implant loading, and one taken in the following 10 years for PES analysis. The radiographs were divided into 4 groups: (1) implant placement; (2) 1-2 years follow-up (short-term); (3) 3-6 years follow-up (medium-term); (4) ≥7 years follow-up (long-term). Photographs were grouped similarly, except that the first group was relative to the day of prosthetic loading. MBL was measured using ImageJ software. Results were analyzed with Generalized Estimating Equations method using SPSS software, the P value was set at <0.05 for significance.

DETAILED DESCRIPTION:
Modern implantology has evolved over the past decades toward solutions that optimize not only the **functional stability** of implants but also the **aesthetic outcome** and the preservation of **hard and soft tissues**. One such innovation is the *convergent transmucosal profile*, a design configuration for dental implants aimed at promoting the coronal migration of collagen fibers, reducing **marginal bone loss (MBL)**, and improving the stability of soft tissues.

**Marginal Bone Loss (MBL)** is a key parameter in assessing the long-term stability of implants and is measured as a reduction in the height of the marginal bone around the implant. The **Pink Esthetic Score (PES)**, on the other hand, qualitatively evaluates the aesthetic outcome of the peri-implant soft tissues by considering parameters such as the shape and fullness of the papilla, the contour of the soft tissues, and the color of the mucosa in relation to the prosthesis.

This **retrospective study** aims to evaluate, in a cohort of patients, the effectiveness of the convergent transmucosal profile of dental implants with respect to bone stability and aesthetic outcomes.

**Study Aim** The main objective of the study is to analyze the **long-term stability** of Marginal Bone Level (MBL) and the Pink Esthetic Score (PES) in a retrospective cohort of patients treated with implants featuring a convergent transmucosal profile. The study intends to identify correlations between aesthetic parameters and bone stability, also evaluating the clinical implications of this implant design.

**Materials and Methods**

**Study Design** The study will be retrospective, based on the analysis of medical records and radiographic data collected in a standardized manner. Selected patients received at least one implant with a convergent transmucosal profile and were followed for **at least 10 years**.

**Inclusion Criteria**

* Adult patients aged between 18 and 75 years.
* Presence of at least one periapical radiograph taken at the time of implant placement and another at 1-2 years, 3-6 years, and 7-10 years after insertion.
* Photographic documentation for PES assessments performed at prosthetic loading and during follow-ups.

**Exclusion Criteria**

* Patients with uncompensated systemic diseases (uncontrolled diabetes, severe autoimmune diseases).
* Heavy smokers (>10 cigarettes per day).
* Incomplete clinical and radiographic documentation.

**Description of the Convergent Transmucosal Profile** The convergent transmucosal profile is characterized by a design that reduces the bulk of the implant neck near the soft tissues. This configuration promotes the coronal migration of collagen fibers, creating a biological seal that helps preserve the bone margin and support the soft tissues, thereby improving aesthetic outcomes.

**Data Collection**

1. **MBL Measurement:** Marginal Bone Loss will be measured using standardized periapical radiographs, with dedicated software such as ImageJ, assessing the distance between the edge of the implant platform and the first bone contact.
2. **PES Evaluation:** The Pink Esthetic Score will be calculated by analyzing photographic images, considering parameters such as the fullness and shape of the papillae, the contour of the soft tissues, mucosal color, and the overall aesthetic integration.

**Sample Size Calculation** The sample size was calculated assuming a clinically relevant difference of 0.5 mm in MBL with a standard deviation of 0.3 mm. With a significance level of 5% and a power of 80%, at least 45 subjects are required. To account for possible dropouts during follow-up, the sample will be increased by 20%, bringing the minimum number to 54 patients.

**Statistical Analysis** Data will be analyzed using SPSS software. Continuous variables will be expressed as means and standard deviations. The data analysis will be conducted using Generalized Estimating Equations (GEE) to manage the dependence between repeated measurements over time. The correlation between MBL and PES will be assessed using the Pearson coefficient. A p-value less than 0.05 will be considered significant.

**Ethical Considerations** The study will be conducted in accordance with the Declaration of Helsinki. All clinical and radiographic data will be anonymized to ensure patient privacy. No additional interventions are planned, and the study does not pose risks to participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 75 years.
* Presence of at least one periapical radiograph taken at the time of implant placement and another at 1-2 years, 3-6 years, and 7-10 years after insertion.
* Photographic documentation for PES assessments performed at prosthetic loading and during follow-ups.

Exclusion Criteria:

* Patients with uncompensated systemic diseases (uncontrolled diabetes, severe autoimmune diseases).
* Heavy smokers (>10 cigarettes per day).
* Incomplete clinical and radiographic documentation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received at least one implant with transmucosal convergent profile
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Marginal bone level | 1 to 10 years after implant placement compared to baseline
  The level of the peri-implant marginal bone measured on intraoral radiograph at various time points
Pink Esthetic Score | from baseline (implant placement) to 10 years
  A scoring system that evaluates the esthetic appearance of soft tissue around dental implants based on five parameters-mesial papilla, distal papilla, curvature and level of facial mucosa, and root convexity/soft-tissue color and texture-each scored from 0 to 2, for a maximum of 10 points

CONTACTS AND LOCATIONS:
Locations (1):
- Cagliari University Hospital, Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No